CLINICAL TRIAL: NCT06149091
Title: Control of Iatrogenic Endobronchial Bleeding by Tranexamic Acid，Adrenalin and Hemagglutinase: a Double-blind Randomized Controlled Trial
Brief Title: Control of Iatrogenic Endobronchial Bleeding by Tranexamic Acid, Adrenalin and Hemagglutinase
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Collaborators: The Second Affiliated Hospital of Harbin Medical University (Other); The First Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Gang Hou, Principal Investigator, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZRJY2021-BJ08-02-01
Record Dates: First submitted 2023-11-20; First posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Iatrogenic Endobronchial Bleeding
Keywords: flexible bronchoscopy; diagnostic flexible bronchoscopy; hemocoagulase; Tranexamic Acid; Adrenalin
MeSH Terms: interventions — Tranexamic Acid; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tranexamic Acid Group (Active Comparator): Patients with iatrogenic airway bleeding who were randomly assigned to the group and failed to achieve hemostasis after three applications of cold saline within a given week were treated with tranexamic acid for hemostasis.
  Interventions: Drug: Tranexamic Acid；
- Adrenalin Group (Active Comparator): Patients with iatrogenic airway bleeding who were randomly assigned to the group and failed to achieve hemostasis after three applications of cold saline within a given week were treated with Adrenalin for hemostasis.
  Interventions: Drug: Adrenalin
- Hemagglutinase Group (Experimental): Patients with iatrogenic airway bleeding who were randomly assigned to the group and failed to achieve hemostasis after three applications of cold saline within a given week were treated with Hemagglutinase for hemostasis.
  Interventions: Drug: Hemagglutinase

INTERVENTIONS:
Drug: Tranexamic Acid； — Tranexamic acid (TXA) is an antifibrinolytic drug that competitively inhibits the activation of plasminogen. After its efficacy and safety were confirmed in several randomized controlled trials, both systemic and topical administration of TXA have been widely used for hemostasis in trauma and various surgical settings.
  Arms: Tranexamic Acid Group
Drug: Adrenalin — In diagnostic bronchoscopy, one of the most commonly used topical hemostatic agent is epinephrine. The primary mechanism of epinephrine is vasoconstriction, leading to reduced blood flow and hemostasis.
  Arms: Adrenalin Group
Drug: Hemagglutinase — Thrombin injection (Batroxobin) is an enzymatic hemostatic agent refined from the venom of the Brazilian lancehead snake. It promotes clot formation at the bleeding site, characterized by rapid and effective hemostasis and high safety. It is now widely used for clinical prevention and treatment of perioperative bleeding and oozing. Multiple randomized controlled studies have evaluated the safety and efficacy of intravenous/topical application of thrombin in various trauma and surgical settings.
  Arms: Hemagglutinase Group

SUMMARY:
A prospective national multi-center study will be conducted to evaluate the effectiveness of hemocoagulase in iatrogenic airway bleeding in a large class III hospital, such as the Second Affiliated Hospital of Harbin Medical University, the First Affiliated Hospital of Nanchang University, and to compare it with topical epinephrine and tranexamic acid in a prospective double-blind cluster randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* During diagnostic bronchoscopy, patients with bronchial bleeding that was not successfully controlled with cold (4°C) saline (3 times within 60 seconds, 5ml each time).

Exclusion Criteria:

* 1: Patients with contraindications for diagnostic flexible bronchoscopy.

  2: Coagulopathy (PV INR >1.3).

  3: Thrombocytopenia (<50x10^9) or anemia (hgb <80 g/L).

  4: Direct oral anticoagulant, low molecular weight heparin, or antiplatelet therapy.

  5: Thrombophilia, history of pulmonary embolism or deep vein thrombosis.

  6: Contraindications for the use of epinephrine in the bronchus.

  7: Coronary artery disease, cerebrovascular disease, history of rapid arrhythmias.

  8: Uncontrolled pulmonary hypertension.

  9: Cardiovascular decompensation.

  10: Severe hypoxia (PaO2 <60mmHg, SaO2 <90%, FiO2 >=60%).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Intratracheal bleeding control rate | Up to a single examination, no more than 1 minute after each drug application. Under bronchoscopy, physicians visually assess clot formation to evaluate bleeding control
  The percentage of iatrogenic bronchial bleeding successfully controlled in each group (%)

SECONDARY OUTCOMES:
Number of tranexamic acid/adrenaline/thrombin applications required to control bronchial bleeding | Until the end of a single procedure (bronchoscopy), up to 1 minute after each drug application.
  Number of tranexamic acid/adrenaline/thrombin applications required to control bronchial bleeding
Number of recurrent bleeding episodes after infusion of tranexamic acid/adrenaline/thrombin (N) | Within 24 hours after a single procedure (bronchoscopy)
  Number of recurrent bleeding episodes after infusion of tranexamic acid/adrenaline/thrombin (N)
Percentage (%) of iatrogenic bronchial bleeding successfully controlled in each group in relation to the severity of the bleeding. | Up to the end of a single procedure (bronchoscopy), a maximum of 1 minute after each drug application.
  Percentage (%) of iatrogenic bronchial bleeding successfully controlled in each group in relation to the severity of the bleeding. Bronchoscopic physicians assess using a Visual Analog Scale (VAS) 1-10 (1 very mild - 10 very severe)

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No